CLINICAL TRIAL: NCT05864911
Title: Efficacy and Safety of the Gastric Bypass Stent System on Body Weight and Metabolic Parameters in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Hangzhou Tangji Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingFH20230327
Record Dates: First submitted 2023-04-03; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: The Gastric Bypass Stent System; total weight loss; excess weight loss; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: placement of the Gastric Bypass Stent System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the Gastric Bypass Stent System group (Experimental): all the participants were implanted with the Gastric Bypass Stent System for 12 weeks and followed up for 24 weeks.
  Interventions: Device: the Gastric Bypass Stent System

INTERVENTIONS:
Device: the Gastric Bypass Stent System — The Gastric Bypass Stent System is a newly designed endoscopic duodenal-jejunal bypass liner for the treatment of obesity by Hangzhou Tangji Medical Technology Co., Ltd.. It consists of three main parts: a 60-cm polyethylene sleeve fixed into the duodenal bulb by anchors with barbs, a delivery system and a retrieval system. Compared to the Endobarrier, it has several technical adjustments. First, it improved sleeve materials to provide better barrier properties and reduce the breeding of bacteria resulting in hepatic abscess. Second, the barbs on the anchoring system have been modified to reduce duodenal injury. Third, the delivery and retrieval system have been optimized to eliminate the need of fluoroscopic guidance during implantation and explantation.

SUMMARY:
In this study, the investigators use a novel endoscopic duodenal-jejunal bypass liner-the Gastric Bypass Stent System (Hangzhou Tangji Medical Technology Co., Ltd., China) for the treatment of obesity. The aim of this study is to evaluate the efficacy and safety of this new device on weight loss and obesity-associated metabolic parameters.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm study conducted at the department of gastroenterology, Beijing Friendship Hospital, Capital Medical University in China. In this study, all the participants were implanted with the Gastric Bypass Stent System. The device had an intended implantation time of 12 weeks, and the participants were followed up for 24 weeks. Both the implantation and explantation were conducted under general anesthesia. A liquid diet was required for a week after implantation to reduce the risk of early obstruction or migration. All the participants received an oral proton pump inhibitor twice daily during the implantation and within 4 weeks of removal. Primary outcomes were changes in excess weight loss and total weight loss at 12 and 24 weeks. Secondary outcomes included changes in body weight, body mass index (BMI), insulin resistance, liver enzymes, lipids and uric acid at 12 and 24 weeks, and device safety. At the first visit, baseline demographics, medical history, physical examination and laboratory tests were collected. The subjects were scheduled for follow-up visit at 1, 4, 12, 16 and 24 weeks. At each visit, body weight was measured and symptoms were recorded. Blood and fecal samples were collected to observe the changes of metabolic parameters and also to monitor the adverse effects. A complete blood count, liver function, blood glucose, insulin, HbA1C, lipids, uric acid, amylase, iron tests and fecal occult blood were partially or all measured at each visit. Insulin resistance was assessed by the homeostasis model assessment of insulin resistance (HOMA-IR), a value ≧2.69 was considered as insulin resistance. Elevated ALT or AST was considered as abnormal liver enzymes. Primary outcomes were changes in EWL and TWL at 12 and 24 weeks. Secondary outcomes included changes in body weight, BMI, insulin resistance, liver enzymes, lipids, UA at 12 and 24 weeks, and device safety.Analyses were conducted with IBM SPSS Statistics for Windows, version 22.0 (IBM Corporation , Armonk, NY). Data was reported as mean ± standard deviation (SD) . A p value of <0.05 was considered statistically significant. Analyses of body weight changes between different time points were conducted with a paired sample t test. Analyses of metabolic parameters in the blood were calculated by generalized estimating equations (GEE) because of the existence of missing values.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤60 years;
* Body mass index ( BMI) ≥30 kg/m2;
* American Society of Anesthesiologists( ASA) Physical Status Classification System:I-II.

Exclusion Criteria:

* Weight loss of more than 4.5 kg in the past three months, or taking weight-lowering drugs in the past month;
* Taking non-steroidal anti-inflammatory drugs (NSAIDs) or antiplatelet drugs or anticoagulant therapy in the past month;
* Previous diagnosis with type 1 diabetes mellitus;
* Loss of islet β-cell function, C-peptide ≤ 1/2 of the normal low limit, or low C-peptide release curve under glucose load;
* Iron deficiency or iron deficiency anemia;
* Severe organ dysfunction of the heart, the lung, the liver or the kidney;
* Patients who have undergone endoscopic retrograde cholangiopancreatography, or have a history of cholecystitis, gallstones with clinical symptoms or stones larger than 20 mm in diameter; pancreatitis or hepatic abscess;
* History of duodenal ulcer or gastric ulcer;
* Patients with gastrointestinal bleeding or potential bleeding;
* Digestive tract malformation, such as digestive tract atresia or previous gastrointestinal surgery that could cause failure of implantation or affect functioning of the device;
* History of intestinal obstruction in the past year;
* Thyroid dysfunction;
* History of systemic lupus erythematosus or scleroderma;
* Pregnant women or women desiring pregnancy in the next few months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline excess weight loss at 4 weeks | 4 weeks
  excess weight loss change
Change from baseline excess weight loss at 12 weeks | 12 weeks
  excess weight loss change
Change from baseline excess weight loss at 24 weeks | 24 weeks
  excess weight loss change
Change from baseline total weight loss at 4 weeks | 4 weeks
  total weight loss change
Change from baseline total weight loss at 12 weeks | 12 weeks
  total weight loss change
Change from baseline total weight loss at 24 weeks | 24 weeks
  total weight loss change
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | within 24 weeks
  Number of participants with treatment-related adverse events to assess device safety

SECONDARY OUTCOMES:
Change from baseline body weight at 4 weeks | 4 weeks
  body weight change
Change from baseline body weight at 12 weeks | 12 weeks
  body weight change
Change from baseline body weight at 24 weeks | 24 weeks
  body weight change
Change from baseline body mass index at 4 weeks | 4 weeks
  body mass index change
Change from baseline body mass index at 12 weeks | 12 weeks
  body mass index change
Change from baseline body mass index at 24 weeks | 24 weeks
  body mass index change
Value change of homeostasis model assessment of insulin resistance at 4 weeks compared with baseline | 4 weeks
  the homeostasis model assessment of insulin resistance were calculated by [fasting insulin level (uU/mL)]×[fasting glucose level (mmol/L)]/22.5
Value change of homeostasis model assessment of insulin resistance at 12 weeks compared with baseline | 12 weeks
  the homeostasis model assessment of insulin resistance were calculated by [fasting insulin level (uU/mL)]×[fasting glucose level (mmol/L)]/22.5
Value change of homeostasis model assessment of insulin resistance at 24 weeks compared with baseline | 24 weeks
  the homeostasis model assessment of insulin resistance were calculated by [fasting insulin level (uU/mL)]×[fasting glucose level (mmol/L)]/22.5
Value change of alanine aminotransferase at 4 weeks compared with baseline | 4 weeks
  value change of alanine aminotransferase
Value change of alanine aminotransferase at 12 weeks compared with baseline | 12 weeks
  value change of alanine aminotransferase
Value change of alanine aminotransferase at 24 weeks compared with baseline | 24 weeks
  value change of alanine aminotransferase
Value change of aspartate aminotransferase at 4 weeks compared with baseline | 4 weeks
  value change of aspartate aminotransferase
Value change of aspartate aminotransferase at 12 weeks compared with baseline | 12 weeks
  value change of aspartate aminotransferase
Value change of aspartate aminotransferase at 24 weeks compared with baseline | 24 weeks
  value change of aspartate aminotransferase
Value change of total cholesterol at 4 weeks compared with baseline | 4 weeks
  value change of total cholesterol
Value change of total cholesterol at 12 weeks compared with baseline | 12 weeks
  value change of total cholesterol
Value change of total cholesterol at 24 weeks compared with baseline | 24 weeks
  value change of total cholesterol
Value change of low density lipoprotein cholesterol at 4 weeks compared with baseline | 4 weeks
  value change of low density lipoprotein cholesterol
Value change of low density lipoprotein cholesterol at 12 weeks compared with baseline | 12 weeks
  value change of low density lipoprotein cholesterol
Value change of low density lipoprotein cholesterol at 24 weeks compared with baseline | 24 weeks
  value change of low density lipoprotein cholesterol
Value change of high density lipoprotein cholesterol at 4 weeks compared with baseline | 4 weeks
  value change of high density lipoprotein cholesterol
Value change of high density lipoprotein cholesterol at 12 weeks compared with baseline | 12 weeks
  value change of high density lipoprotein cholesterol
Value change of high density lipoprotein cholesterol at 24 weeks compared with baseline | 24 weeks
  value change of high density lipoprotein cholesterol
Value change of triglyceride at 4 weeks compared with baseline | 4 weeks
  value change of triglyceride
Value change of triglyceride at 12 weeks compared with baseline | 12 weeks
  value change of triglyceride
Value change of triglyceride at 24 weeks compared with baseline | 24 weeks
  value change of triglyceride
Value change of blood uric acid at 4 weeks compared with baseline | 4 weeks
  value change of blood uric acid
Value change of blood uric acid at 12 weeks compared with baseline | 12 weeks
  value change of blood uric acid
Value change of blood uric acid at 24 weeks compared with baseline | 24 weeks
  value change of blood uric acid

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The baseline demographics, the body weight changes，blood and fecal tests at each visit and the adverse effects will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available after half a year and for 3 years.
Access Criteria: all the researcher interested can get access.

REFERENCES:
- [Background] Wang L, Zhou B, Zhao Z, Yang L, Zhang M, Jiang Y, Li Y, Zhou M, Wang L, Huang Z, Zhang X, Zhao L, Yu D, Li C, Ezzati M, Chen Z, Wu J, Ding G, Li X. Body-mass index and obesity in urban and rural China: findings from consecutive nationally representative surveys during 2004-18. Lancet. 2021 Jul 3;398(10294):53-63. doi: 10.1016/S0140-6736(21)00798-4. PMID 34217401
- [Background] India State-Level Disease Burden Initiative CVD Collaborators. The changing patterns of cardiovascular diseases and their risk factors in the states of India: the Global Burden of Disease Study 1990-2016. Lancet Glob Health. 2018 Dec;6(12):e1339-e1351. doi: 10.1016/S2214-109X(18)30407-8. Epub 2018 Sep 12. PMID 30219317
- [Background] Ren M, Zhou X, Yu M, Cao Y, Xu C, Yu C, Ji F. Prospective study of a new endoscopic duodenal-jejunal bypass sleeve in obese patients with nonalcoholic fatty liver disease (with video). Dig Endosc. 2023 Jan;35(1):58-66. doi: 10.1111/den.14409. Epub 2022 Aug 23. PMID 35869797